CLINICAL TRIAL: NCT06283472
Title: Enhancing Prospective Thinking in Early Recovery
Brief Title: Enhancing Prospective Thinking in Early Recovery (BEAM)
Acronym: BEAM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Brandon G. Oberlin, PhD, Assistant Professor, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1805574553; Aims 14-16; 2P60AA007611-403343 (Other Grant/Funding Number: National Institute on Alcohol Abuse and Alcoholism); 2P60AA007611 (NIH)
Record Dates: First submitted 2024-02-21; First posted 2024-02-28 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Alcohol Use Disorder
Keywords: Alcohol Use Disorder; Alcohol Abuse; Heavy Drinking; Alcohol
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Who Masked: Participant
Masking Description: Eligible participants will be randomly assigned to either the high-intensity (experimental) or low-intensity (control) groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High-Intensity (Experimental): Participants will receive high-intensity episodic future-thinking cue images, and high-intensity episodic recent-thinking cue images during an MRI decision-making task.
  Interventions: Behavioral: High-Intensity Cue
- Low-Intensity (Control) (Active Comparator): Participants will receive low-intensity episodic future-thinking cue images, and low-intensity episodic recent-thinking cue images during an MRI decision-making task.
  Interventions: Behavioral: Low-Intensity Cue

INTERVENTIONS:
Behavioral: High-Intensity Cue — Participants in the high-intensity group will receive high-intensity image cues that represent self-reported events they did on the previous day and self-reported events they look forward to in the future.
  Arms: High-Intensity
Behavioral: Low-Intensity Cue — Participants in the low-intensity group will receive low-intensity image cues that represent self-reported events they did on the previous day and self-reported events they look forward to in the future.
  Arms: Low-Intensity (Control)

SUMMARY:
The goal of this clinical trial is to test the prosocial effects of personally-relevant, high-intensity episodic future-thinking (EFT) cues in alcohol use disorder persons and related brain mechanisms. The main question[s] this trial aims to answer are:

* Will high-intensity EFT cues will produce greater delayed reward preference than low-intensity cues?
* Will high-intensity EFT cues effect greater treatment-seeking interest?
* Will high-intensity EFT cues elicit greater response in regions for prospective thinking during delay discounting (vs. low-intensity)
* Will nucleus accumbens-precuneus resting connectivity correlate with behavioral SS?
* Will the novel behavioral SS decision-making task activate the nucleus accumbens?

Researchers will compare the experimental (high-intensity group) and control (low-intensity) groups to see if there are differences in the results for the questions outlined above.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who meet current heavy drinking (≥2 heavy drinking days/month OR ≥7 drinks/week for biological females, and ≥14 drinks/week if biological male [NIAAA definition] and/or AUDIT scores ≥8)
* English comprehension

Exclusion Criteria:

* Unstable medical disorders
* Outside the age range of 18-60
* Smell/taste disorders
* Unstable psychiatric conditions

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Estimated)
Dates: Start 2024-06-17 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Increase Prospective Thinking | Study Day Visit (Day 1)
  High-intensity episodic future-thinking image cues will change prospective thinking.
Delayed Rewards | Study Day Visit (Day 1)
  High-intensity episodic future-thinking image cues will change preference for delayed rewards, which will be measured using a behavioral delayed discounting task.

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University School of Medicine - Goodman Hall, Indianapolis, Indiana, United States